CLINICAL TRIAL: NCT06126783
Title: A Multicenter, Open-label Extension Study Evaluating the Efficacy and Safety of IBI311 in Subjects With Thyroid Eye Disease
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI311A301
Record Dates: First submitted 2023-10-19; First posted 2023-11-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Thyroid Eye Disease, TED
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBI311 (Experimental): The first dose was 10 mg/kg, followed by 7 maintenance doses of 20 mg/kg, Q3W
  Interventions: Drug: IBI311

INTERVENTIONS:
Drug: IBI311 — The first dose was 10 mg/kg, followed by 7 maintenance doses of 20 mg/kg, Q3W

SUMMARY:
A multicenter, open-label extension study evaluating the efficacy and safety of IBI311 in subjects with thyroid eye disease

DETAILED DESCRIPTION:
This is a multicenter, open-label outreach study. Participants who have previously participated in and completed CIBI311A201 double-blind treatment can enter this study after signing informed consent. The study included an observation period and an open treatment period. Observation period: From weeks D0 to 24, all subjects will return to the research center every 8 weeks for disease evaluation. If the investigator determines that treatment is required based on predefined criteria, they will enter the open treatment period to receive IBI311 treatment; Otherwise, subjects will continue to be visited every 8 weeks until week 24. Open Treatment period: Subjects entering the open treatment period will receive 8 infusions of IBI311 (initial dose of 10 mg/kg, followed by 7 maintenance doses of 20 mg/kg, Q3W.

ELIGIBILITY:
Inclusion Criteria:

1. Comply with the test procedure and voluntarily sign the informed consent;
2. Male or female subjects aged between 18 and 80 years (inclusive) at the time of FU1 visit;
3. For subjects who completed CIBI311A201 double-blind treatment period, the cohort date from the end of CIBI311A201 study was no more than 28 days;
4. If the subject is female, it should be postmenopausal or after surgical sterilization or FU1 visit urine pregnancy test negative and agree to take contraceptive measures within 120 days from FU1 visit to the last dose Women of childbearing age; Male subjects should agree to use contraception within 120 days from the FU1 visit to the last dose.

Exclusion Criteria:

1. Visual dysfunction due to optic neuropathy, defined as a decrease of ≥2 lines of best corrected vision within the last 180 days, a new visual field defect, or color difference secondary to optic nerve involvementOften;
2. Patients with corneal ulcers that the investigator determined did not resolve after treatment;
3. When the FU1 visit predecessor was scheduled to receive orbital radiation therapy or surgery for TED, including orbital decompression, strabismus correction, and eyelid correction, or during the study periodEtc.;
4. Poor thyroid function control was defined as free T3 or T4 deviating from the normal reference range of the local research center laboratory by more than 50% during FU1 visit;
5. The presence of any other prior disease, metabolic disorder, abnormal results of physical examination or clinical laboratory examination, which may reasonably be suspected to cause contraindications in the use of the test drug, or shadow Diseases or conditions that place subjects at high risk for treatment complications, including, but not limited to, confirmed or clinically suspected inflammatory bowel disease and coagulation Blood dysfunction, history of acute cardiovascular and cerebrovascular disease or treatment within 180 days prior to FU1 visit (including but not limited to: cerebrovascular accident, transient cerebral ischemia, acute myocardial infarction) Death, unstable angina pectoris, coronary artery bypass grafting, percutaneous coronary intervention (except diagnostic angiography), severe arrhythmia, etc.), treatment within the past 5 years or A history of untreated malignancy (squamous cell carcinoma of the skin, basal cell carcinoma, carcinoma in situ of the cervix, prostate in situ, or thyroid that has been successfully resected without evidence of metastasis) Other than papillary carcinoma), serious systemic infection, non-TED caused eye protrusion, etc.;
6. At the time of FU1 visit, either ear was present: a history of tinnitus or other hearing impairment; Or abnormal pure tone audiometry (defined as 0.5 1 24 4 kHz mean bone conduction threshold ≥25 dB or either Bone conduction threshold under frequency ≥40 dB);
7. When FU1 visited, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) were 3 times higher than ULN;
8. When FU1 was visited, Glomerular Filtration Rate (GFR) was < 30 ml/min/1.73 m2 (MDRD formula: GFR =186× serum creatinine (mg/dl)).-1.154× (age) -0.203× (0.742 [if female]), unit conversion of blood creatinine: 1 μmol/L=0.0113 mg/dL);
9. The presence of poorly controlled diabetes at FU1 visit (defined as ≥9.0% HBA1C at FU1 visit or a new diabetes medication within 60 days prior to screening]Dose change of diabetes drugs currently prescribed > 10%);
10. At FU1 visit, poorly controlled hypertension was present, with systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg; Or FU1 adjusted blood pressure medication (dose or.) within 30 days prior to visit Type of drug); Renal artery stenosis; Or evidence of unstable blood pressure (including postural hypotension);
11. A 12-lead ECG showing a heart rate < 50 beats/min or > 100 beats/min at the FU1 visit indicates active heart disease, or an ECG abnormality at the time of the FU1 visit, as the investigator believes Interfering with the interpretation of ECG results during follow-up, especially excluding QTcF > 500 ms;
12. Subjects received systemic or local use of glucocorticoids, immunosuppressants, or biologics (CD20 antibody, interleukin) from the end of CIBI311A201 study until FU1 visit of this study-6 receptor antibody, tetulizumab, etc.) to treat TED;
13. Subjects treated TED with selenium or biotin (except multivitamins containing selenium or biotin) from the end of CIBI311A201 study to before FU1 visit of this study;
14. Subjects had participated in other interventionary clinical trials (e.g., for drugs, during their 5 half-lives, with older participants) from the end of the CIBI311A201 study until the FU1 visit of this study Allowed; Vitamins and minerals), or attempting to participate in other clinical trials during the study period;
15. Pregnant and lactating female subjects;
16. People who are known to be allergic to the ingredients of the investigational drug, or have a pre-existing allergy to other monoclonal antibodies;
17. Participants considered unsuitable for this clinical trial due to other reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The response rate of exophthalmos was studied. | After receiving IBI311 treatment for 24 weeks
  To evaluate the effect of IBI311 on the exophthalmos response rate in the study eye (defined as the percentage of subjects with an exophthalmos reduction of ≥2 mm from baseline in the study eye without an increase of ≥2 mm in the contralaterial eye).

SECONDARY OUTCOMES:
Overall responder rate (i.e., percentage of subjects with a ≥ 2-point decrease in Clinical Activity Score [CAS] and a ≥ 2 mm decrease from baseline in proptosis in the study eye, and without corresponding deterioration in the fellow eye in the study eye | After receiving IBI311 treatment for 24 weeks
  Total ocular response rate in the study eyes after 4 /8 IBI311 treatments.
To evaluate the effects of IBI311 on ocular CAS score. | After receiving IBI311 treatment for 24 weeks
  Percentage of subjects with a CAS value of 0 or 1 after 4 /8 IBI311 treatments.
To evaluate the effects of IBI311 on exophthalmos. | After receiving IBI311 treatment for 24 weeks
  Mean change in exophthalmia from baseline in study eyes after 4 /8 IBI311 treatments.Efficacy of investigational eye therapy after 4 /8 IBI311 treatments
To evaluate the efficacy of IBI311 in improving contralateral eye. | After receiving IBI311 treatment for 24 weeks
  After 4 /8 treatments with IBI311,The response rate of exophthalmos in the improving contralateral eye.
To evaluate the efficacy of IBI311 in improving diplopia. | After receiving IBI311 treatment for 24 weeks
  Diplopia response rate after four/eight IBI311 treatments (defined as the percentage of subjects with diplopia at baseline with grade 1 reduction).
To evaluate the effects of IBI311 on Graves' ophthalmopathy-specificquality of life (GO-QOL) scores. | After receiving IBI311 treatment for 24 weeks
  Mean change in total GO-QOL questionnaire scores from baseline after 4/8 IBI311 treatments；
The rate of TED recurrence after discontinuation of IBI311 treatment was assessed | After receiving IBI311 treatment for 24 weeks
  Proportion of subjects entering open treatment due to relapse.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | After receiving IBI311 treatment for 24 weeks
  Incidence, association with the study drug and severity of ocular and systemic adverse events (AE), treatment-emergent adverse events (TEAE), and serious adverse events (SAE)

CONTACTS AND LOCATIONS:
Locations (1):
- Ninth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China